CLINICAL TRIAL: NCT02675504
Title: Validation of a Scale of Self-assessment of Fear Faces in Children 4 to 12 Years: Scary Scale
Brief Title: Validation of a Scale of Self-assessment of Fear Faces in Children 4 to 12 Years
Acronym: TROUILLOMETRE
Status: Completed | Type: Observational
Sponsor: University Hospital, Limoges (Other)
Responsible Party: Sponsor
Other Study IDs: I14006
Record Dates: First submitted 2016-02-03; First posted 2016-02-05 (Estimated); Last update posted 2019-01-11 (Actual); Status verified 2016-03

CONDITIONS: Fear
Keywords: scary scale

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: Placing a scale self-assessment of fear — Children spend a self-assessment scale of fear

SUMMARY:
Since the 2000s, the experiences of children and especially their fear during a consultation, a treatment or examination is food for thought in our establishment. There is no tool validated self-assessment of fear to 6 faces. It therefore appeared necessary to us to create this tool. The scale self-assessment of the fear that we have developed consists of six faces representing a gradual level of fear: the child can easily describe their level of fear, which allows for appropriate care.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 4 to 12 years.
* Enrolled in one of the participating institutions in the study (steps 1-5) or consultant pediatric emergencies at the Children of Limoges (step 6).
* Authorization of at least one person having parental authority for the child to participate in the study.
* Children affiliates or benefiting from a social security

Exclusion Criteria:

* Children with psychomotor disorders that prevent the use of the scale studied and understanding instructions.
* Children in vital emergency

Ages: 4 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Participating in the study of children aged 4 to 12 years. In this study, participation of school children and hospitalized children
Sampling Method: Probability Sample
Enrollment: 544 (Actual)
Dates: Start 2016-03 (Actual); Primary Completion 2016-10 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Percentage of children who validate the 6 faces expressing fear. | 5 minutes
  Percentage of children who validate the 6 faces expressing fear. The test will be validated if we get a result at least 60%.

SECONDARY OUTCOMES:
Percentage of children who properly fit the faces expressing fear in ascending and descending order. | 5 minutes

CONTACTS AND LOCATIONS:
Locations (1):
- Limoges hospital, Limoges, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Thurillet S, Bahans C, Wood C, Bougnard S, Labrunie A, Messager V, Toniolo J, Beloni P, Fourcade L. Psychometric properties of a self-assessment fear scale in children aged 4 to 12 years. Scary Scale. J Pediatr Nurs. 2022 Jul-Aug;65:108-115. doi: 10.1016/j.pedn.2022.02.020. Epub 2022 Mar 14. PMID 35300885